CLINICAL TRIAL: NCT03403244
Title: US-MR Image Fusion-guided Versus Fluoroscopy-guided Percutaneous Transforaminal Endoscopic Discectomy for the Treatment of Lumbar Disc Herniation: a Comparative Cohort Study
Brief Title: US-MR Image Fusion-guided Percutaneous Transforaminal Endoscopic Discectomy for the Treatment of Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Limin Rong, proffesor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US-MR guided PTED for LDH
Record Dates: First submitted 2018-01-04; First posted 2018-01-18 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Lumbar Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-MR image fusion-guided PTED (Experimental): US-MR image fusion-guided PTED: the puncture procedure during PTED was performed under the guidance of ultrasound-MR fusion technique.
  Interventions: Procedure: US-MR image fusion-guided PTED
- fluoroscopy-guided PTED (Active Comparator): fluoroscopy-guided PTED: the puncture procedure during PTED was performed under the guidance of fluoroscopy.
  Interventions: Procedure: fluoroscopy-guided PTED

INTERVENTIONS:
Procedure: US-MR image fusion-guided PTED — patients diagnosed with lumbar disc herniation undergoing US-MR image fusion-guided PTED
  Arms: US-MR image fusion-guided PTED
Procedure: fluoroscopy-guided PTED — patients diagnosed with lumbar disc herniation undergoing fluoroscopy-guided PTED
  Arms: fluoroscopy-guided PTED

SUMMARY:
The purpose of this study is to evaluate the feasibility and efficacy of US-MR image fusion-guided percutaneous transforaminal endoscopic discectomy for the treatment of lumbar disc herniation

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common pathological process leading to spinal surgery. Open discectomy used to be a widespread procedure for surgical treatment for symptomatic LDH. Currently, with rapid progress of endoscopic techniques, several minimal invasive endoscopic surgeries have been developed to perform discectomy. Percutaneous transforaminal endoscopic discectomy (PTED) a widely used minimal invasive surgical procedures, the effectiveness of which has been proved to be comparable to conventional open discectomy. However, the use of fluoroscopy may be usually required to indirectly visualize pertinent anatomy to achieve an optimal result on radiographs. As we known, increased radiation exposure may be associated with potential stochastic and deterministic adverse events. Therefore, it is important to reduce the radiation dose of practitioners to minimize risk of potential radiation-induced complications.

Ultrasound-MR fusion technique combines the advantages of ultrasound and MR, and overcome the shortcomings of each single imaging method. It provides MR cross-sectional multiplanar images that correspond to the acquired real-time US images, and all images can be displayed simultaneously and in real time according to the angle of the US transducer. US-MR fusion image has been widely used in prostate and liver intervention. However, to our limited knowledge, there is only one research about the application of US-MR fusion image in lumbar spinal surgery.

In this study, a comparative cohort study will be performed to evaluate feasibility and efficacy of US-MR image fusion-guided percutaneous transforaminal endoscopic discectomy for the treatment of lumbar disc herniation(LDH). We will conduct the study at the 3rd affiliated hospitals of Sun Yat-Sen University.

Two groups of patients will be investigated: patients diagnosed with lumbar disc herniation undergoing US-MR image fusion-guided PTED (US-MR PTED), and fluoroscopy-guided PTED (FL PTED).

The primary outcomes of the study will be radiation exposure and puncture time. Secondary outcomes include fusion efficacy, puncture accuracy, puncture satisfaction of surgeon, comfort of patient and clinical effectiveness.

On the basis of the results of this trial we will, for the first time, have scientific evidence as to the feasibility and efficacy of US-MR image fusion-guided percutaneous transforaminal endoscopic discectomy for the treatment of lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

1. persistent radicular pain.
2. an imaging study (MRI or CT) showing LDH at a level and side corresponding to the patient
3. single responsible segment of lumbar disc herniation
4. L4-5 segment

Exclusion Criteria:

1. Cauda equina syndrome or progressive neurologic deficit requiring urgent surgical intervention
2. Combination with other spinal disorder requiring advanced surgery (such as lumbar stenosis, spondylolisthesis, deformity, fracture, infection, tumor and so on)
3. Equal to or more than two responsible level
4. Previous spinal surgery
5. unable to collaborate during surgery
6. far-lateral disc herniation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
radiation exposure | during operation
  dose of radiation exposure

SECONDARY OUTCOMES:
puncture accuracy | during operation
  the accuracy of puncture position confirmed by fluoroscopy.
puncture satisfaction of surgeon | during operation
  use Visual Analog Scales (VAS,scores ranging from 0 to 10, with higher scores indicating more satisfactory) to evaluate the satisfaction of surgeon during puncture
comfort of patient | during operation
  use Visual Analog Scales (VAS,scores ranging from 0 to 10, with higher scores indicating more comfortable) to evaluate the comfort of patient during puncture
degree of pain | preoperation, immediately postoperation, 1 week postoperation
  Visual Analog Scales (VAS, scores ranging from 0 to 10, with higher scores indicating more severe pain)
degree of disability | preoperation, immediately postoperation, 1 week postoperation
  Oswestry Disability Index (ODI) score (ranging from 0 to 100, with higher scores indicating more disability related to pain）
puncture time | during operation
  the time from the begin of puncture to the confirmation of optimal puncture

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xie P, Feng F, Cao J, Chen Z, He B, Kang Z, He L, Wu W, Tan L, Li K, Zheng R, Rong L. Real-time ultrasonography-magnetic resonance image fusion navigation for percutaneous transforaminal endoscopic discectomy. J Neurosurg Spine. 2020 Mar 27;33(2):192-198. doi: 10.3171/2020.1.SPINE191223. Print 2020 Aug 1. PMID 32217792